CLINICAL TRIAL: NCT06978725
Title: A Phase 2 Randomized, Double-Blind, Placebo-Controlled, Dose-Ranging Study to Investigate the Safety and Efficacy of Oral Brepocitinib in Adults With Cutaneous Sarcoidosis
Brief Title: A Phase 2 Study of the Safety and Efficacy of Brepocitinib in Adults With Cutaneous Sarcoidosis (BEACON)
Acronym: BEACON
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Priovant Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PVT-2201-203
Record Dates: First submitted 2025-04-30; First posted 2025-05-18 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Cutaneous Sarcoidosis
Keywords: sarcoidosis; cutaneous sarcoidosis; brepocitinib
MeSH Terms: conditions — Sarcoidosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Brepocitinib Dose Level 1 (Experimental)
  Interventions: Drug: Oral Brepocitinib
- Brepocitinib Dose Level 2 (Experimental)
  Interventions: Drug: Oral Brepocitinib
- Placebo (Placebo Comparator)
  Interventions: Drug: Oral Placebo

INTERVENTIONS:
Drug: Oral Brepocitinib — Drug: Oral Brepocitinib
  Arms: Brepocitinib Dose Level 1; Brepocitinib Dose Level 2
Drug: Oral Placebo — Drug: Oral Placebo
  Arms: Placebo

SUMMARY:
This study will evaluate the clinical safety and efficacy of oral brepocitinib in participants with cutaneous sarcoidosis.

ELIGIBILITY:
Inclusion Criteria:

1. Adults subjects (18-74)
2. Cutaneous sarcoidosis with characteristic skin biopsy histology
3. A CSAMI activity score ≥ 10
4. Weight > 40 kg to < 130 kg with BMI < 40 kg/m2 .

Exclusion Criteria

1. History of

   * Lymphoproliferative disorder
   * Active malignancy;
   * History of cancer within 5 years prior to baseline (exceptions for basal cell carcinoma, squamous cell carcinoma, or carcinoma in situ of the uterine cervix).
2. High risk of thrombosis or cardiovascular disease
3. High risk of herpes zoster
4. Active or recent infection

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2025-04-09 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Treatment Emergent Adverse Events and Serious Adverse Events as assessed by CTCAE v5.0 | Screening up to 28 days after the last dose of study drug at 16 weeks

SECONDARY OUTCOMES:
Change from baseline in the Cutaneous Sarcoidosis Activity and Morphology Instrument Activity (CSAMI-A) score through Week 16. | 16 Weeks
  CSAMI-A score is a measure of cutaneous sarcoidosis disease activity. A higher score indicates worse disease. Scores range from 0-165.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Clinical Trial Site, San Francisco, California
  - Clinical Trial Site, Durham, North Carolina
  - Clinical Trial Site, Philadelphia, Pennsylvania
  - Clinical Trial Site, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided